CLINICAL TRIAL: NCT01869751
Title: The Colonic Transit Time: a Modifiable Determinant of Intestinal Production and Uptake of Microbial Metabolites?
Status: Withdrawn | Type: Observational
Why Stopped: failure to recruit patients
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S55296
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prucalopride: Slow-transit constipation with treatment with prucalopride
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: Prucalopride — Treatment with prucalopride for slow-transit constipation

SUMMARY:
Chronic kidney disease is associated with the accumulation of various metabolites, i.e., uremic retention solutes. Evidence is mounting that the colonic microbiome contributes substantially to these uremic retention solutes. Indoxyl sulfate and p-cresyl sulfate are among the most extensively studied gut microbial metabolites, and are associated with cardiovascular disease, chronic kidney disease progression and overall mortality. Colonic transit time is an important determinant of intestinal generation and uptake of bacterial metabolites. However, it is unknown if accelerating the colonic transit time reduces the intestinal generation and uptake of indoxyl sulfate and p-cresyl sulfate. Prucalopride is a selective, high-affinity 5-HT4 receptor agonist with a stimulating effect on colonic motility and transit. It is currently used in treating chronic slow-transit constipation. An observational study will be initiated in non-chronic kidney disease patients with chronic slow-transit constipation necessitating treatment with prucalopride to observe its effect on serum concentrations and intestinal generation of indoxyl sulfate and p-cresyl sulfate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 85 years
* Chronic slow-transit constipation as defined be 4 criteria:

  1. having two or fewer spontaneous complete bowel movements week for a minimum of 6 months
  2. having one or more of the following symptoms for at least one-quarter of the time: lumpy/hard stools, a sensation of incomplete evacuation, or straining during defecation.
  3. slow transit time as determined by Rx colon transit study ("pellet")
  4. without evidence of secondary constipation or primary defecation disorder
* Need of therapy with prucalopride (i.e., inefficacy of dietary changes and laxatives)
* Follow-up visit possible after 4 weeks of treatment
* Written informed consent

Exclusion Criteria:

* History or new diagnosis of organic intestinal disease (e.g., inflammatory bowel disease, malignancy)
* Secondary constipation (drug-induced, endocrine, metabolic or neurological disorders, surgery, known or suspected organic disorders of the large intestine, or megacolon) or primary defecation disorder
* Use of laxatives two days before start of treatment and during treatment period. If there is no spontaneous bowel movement during 3 consecutive days, rescue treatment with bisacodyl and/or enema is allowed if necessary
* Presence of significant co-morbidity (uncontrolled heart, liver and lung disease)
* Pregnancy
* Chronic kidney disease, i.e., estimated glomerular filtration rate (MDRD) < 60 ml/min/m² or need of dialysis therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or newly diagnosed chronic slow-transit constipation necessitating treatment with prucalopride (Resolor®, Shire) according to current treatment guidelines
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
change in serum concentration of bacterial metabolites | 4 weeks
  change in serum concentration of bacterial metabolites before and after (4 weeks) treatment of prucalopride

SECONDARY OUTCOMES:
change in 24h urinary excretion rate of bacterial metabolites | 4 weeks
  change in 24h urinary excretion rate of bacterial metabolites before and after (4 weeks) treatment of prucalopride

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Poesen, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Björn Meijers, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Jan Tack, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium